CLINICAL TRIAL: NCT07374172
Title: SADT in COPD and Oscillometry in Obstructive Airway Disease in Primary Care. The SCOOP-study
Acronym: SCOOP
Status: Active, not recruiting | Type: Observational
Sponsor: General Practitioners Research Institute (Network)
Responsible Party: Sponsor
Other Study IDs: GPRI-2024-002
Record Dates: First submitted 2026-01-15; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Asthma; COPD; Small Airway Disease
Keywords: SADT-c; Oscillometry
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with Small Airway Disease
  Interventions: Diagnostic Test: Oscillometer ALDS
- Participants without Small Airway Disease
  Interventions: Diagnostic Test: Oscillometer ALDS

INTERVENTIONS:
Diagnostic Test: Oscillometer ALDS — Oscillometry is a non-invasive technique for assessing lung function, as it requires only 45-60 seconds of tidal breathing to measure the mechanical properties of the respiratory system. This makes the measurement suitable for patients of all ages and with severe respiratory conditions. It also reduces the number of errors as compared to other methods (e.g., spirometry). Oscillometry can be used to evaluate airway resistance, reactance, and compliance, insights that are challenging to obtain with other methods. This quality makes oscillometry especially sensitive for obstructive diseases like asthma and COPD, and correlations with physiological small airways dysfunction have also been shown
  . The Ambulatory Lung Diagnosis System (ALDS), manufactured by Lothar MedTec, can be used to perform oscillometry and spirometry. The ALDS follows the European Respiratory Society (ERS) technical standards for measurement and reporting of oscillometry.

SUMMARY:
Rationale: The Small Airways are a major site of obstruction in many respiratory diseases, including COPD. More insight into a diagnosis of Small Airways Dysfunction (SAD) in patients with COPD is clinically valuable as it might enable tailored pharmacotherapy. Currently, methods to diagnose SAD in COPD are not standardized and are not available in routine clinical practice. The Small Airways Dysfunction Tool (SADT) was developed to identify patients with asthma and SAD. Initially, the SADT included a comprehensive 63-item questionnaire. The number of items has been reduced to a SADT-asthma (SADT a) questionnaire and key patient and disease characteristics for it to be feasible and implementable in clinical practice. Although there are many similarities between asthma and COPD, there might be differences in clinical characteristics and responses to small airways dysfunction between the two diseases. The current study aims to adapt the original 63-item SADT questionnaire for dedicated use in COPD by reducing the number of items, and identifying COPD-SAD-specific items, to enhance its efficiency in identifying SAD when combined with key patient and disease characteristics in individuals with COPD (SADT-c). In addition, a comparison of diagnostic accuracy of spirometry and oscillometry will be made by interpretations by a panel of experts to provide a triage diagnosis. The previously developed machine learning AC/DC tool will be used to explore its diagnostic accuracy using oscillometry and spirometry results. This can contribute to standardizing oscillometry in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Suspected of having COPD, asthma or ACO as indicated by the referring GP OR a previous diagnosis of COPD

Exclusion Criteria:

* Inability to understand and sign the written informed consent form.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population for the SCOOP study will consist of patients referred by their General Practitioner (GP) to the Asthma/COPD service. Patients can be referred by their GP when they are suspected to have asthma, Chronic Obstructive Pulmonary Disease (COPD), asthma-COPD overlap (ACO) or when they present with pulmonary symptoms of unknown origin. After referral by the GP, patients will be invited by the Asthma/COPD service. Both patients invited for an initial diagnostic visit or a control visit can participate in the SCOOP study.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The predictive value of SADT-c for detecting SAD in patients with COPD. | At baseline study visit, during pulmonary function testing
  To determine whether SADT-c can be used in patients with COPD to detect SAD.

SECONDARY OUTCOMES:
Predictive value of SADT-a bronze model for SAD in COPD. | At baseline study visit, during pulmonary function testing
  To determine whether the bronze model SADT-a is predictive for SAD in COPD.
Develop SADT-c. | At baseline study visit, using data collected during pulmonary function testing and clinical assessment
  Agreement between SADT-c results and disease parameters.
To evaluate how SADT-c compares to SADT-a. | At baseline study visit, during pulmonary function testing
  Relative predictive value of SADT-a versus SADT-c for SAD in COPD defined as R5-R20 > ULN1
To determine whether oscillometry and spirometry are equally effective for triage diagnosis in patients in primary care with respiratory symptoms. | At baseline study visit, during initial diagnostic assessment in primary care
  Agreement between triage diagnoses from oscillometry and spirometry. Relative usability of spirometry and oscillometry.
Assess the diagnostic performance of the Asthma/COPD Differentiation Classification (AC/DC) Tool. | At baseline study visit, with expert panel diagnosis based on data collected during the study assessment
  Diagnostic performance of AC/DC tool compared to expert panel diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Primary care sites across the Netherlands, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No